CLINICAL TRIAL: NCT02781961
Title: Identification of In-vivo Probe Based Confocal Laser Endomicroscopy (pCLE) Gastric & Duodenal Cellular Characteristics in Obese Women Before & After Weight Reduction
Brief Title: Identification of In-vivo Probe Based Confocal Laser Endomicroscopy Cellular Characteristics in Obese Women
Status: Terminated | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ofir Harnoy MD, Dr, Sheba Medical Center
Other Study IDs: SMC-15-2353
Record Dates: First submitted 2016-05-17; First posted 2016-05-25 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: cellvizio — pCLE during gastroscopy

SUMMARY:
Previous studies have shown that histological changes in the gastric mucosa between obese and non-obese individuals do exist. Understanding these histological differences (between obese and non-obese individuals) might elucidate obesity pathophysiology.

However, the data is scarce and even contradictory. Even less is known about the histological characteristics of the duodenal mucosa in obesity and lean states, but several studies already performed hint for some differences. These differences might influence gut hormones composition and function and play a crucial role in the development of obesity and metabolic syndrome. To our best knowledge, in-vivo, human, real-time cellular level comparison of gastric and duodenal mucosa has never been done. This can be now accomplished with pCLE.

pCLE, is composed from a miniature microscope assembled in the tip of an optical fiber. This optic fiber is then inserted through the working channel of a standard endoscope, bringing the microscope at the tip of the fiber to close proximity with the tissue. The system applies a blue-light laser that after staining with fluorescein (IV 2.5 ml, 10% fluorescein, once) provides a cellular-level, in-vivo, real time images: the concept of so called "optical biopsies". The system has been used as an auxiliary tool in GI-endoscopy in recent years. This technology has been shown to be useful in identifying objective histological features and even intramucosal bacteria in different tissues.

DETAILED DESCRIPTION:
Previous studies have shown that histological changes in the gastric mucosa between obese and non-obese individuals do exist, mainly in the cells producing the hormone ghrelin, but also in other gut hormones. Understanding these histological differences (between obese and non-obese individuals) might elucidate obesity pathophysiology, however, the data is scarce and even contradictory. Even less is known about the histological characteristics of the duodenal mucosa in obesity and lean states, but several studies already performed hint for some differences.. In conclusion, the investigators assume that obese and non-obese individuals may have gastric and/or duodenal histological differences. These differences might influence gut hormones composition and function and play a crucial role in the development of obesity and metabolic syndrome. To our best knowledge, in-vivo, human, real-time cellular level comparison of gastric and duodenal mucosa as well as differences in the microbiome of the stomach and duodenum between obese and non-obese individuals has never been done. This can be now accomplished with pCLE.

pCLE, is composed from a miniature microscope assembled in the tip of an optical fiber. This optic fiber is then inserted through the working channel of a standard endoscope, bringing the microscope at the tip of the fiber to close proximity with the tissue. The system applies a blue-light laser that after staining with fluorescein (IV 2.5 ml, 10% fluorescein, once) provides a cellular-level, in-vivo, real time images: the concept of so called "optical biopsies". The system has been used as an auxiliary tool in GI-endoscopy in recent years. This technology has been shown to be useful in identifying objective histological features and even intramucosal bacteria in different tissues.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* BMI>= 35 with MS or
* BMI>=40 without MS

Exclusion Criteria:

* HIV infection
* Active Helicobacter Pylori infection
* CELIAC disease
* Autoimmune gastritis as defined by B12 deficiency and the presence of anti-intrinsic factor/ anti-parietal Ab's
* Concomitant disease with potential upper GI involvement
* Pregnancy
* Participation in another clinical trial
* Declined to sign an informed consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients, referred for bariatric sleeve gastrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-06; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
tissue morphology | 3 months
  pCLE morphological characteristics of gastric and duodenal cells in obese individuals, before and after sleeve gastrectomy (when weight loss is achieved)

CONTACTS AND LOCATIONS:
Overall Officials: OFIR HAR-NOY, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No